CLINICAL TRIAL: NCT06724705
Title: Testing the Capability of the Smart Underwear Device to Detect Increased Microbiome Activity Following Lactose Consumption
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, College Park (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: Smart Underwear Lactose
Record Dates: First submitted 2024-11-25; First posted 2024-12-09 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Lactose Intolerance, Adult Type
MeSH Terms: conditions — Lactose Intolerance, Adult Type | interventions — Lactose; Sucrose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): Participants consume sucrose and wear the Smart Underwear device
  Interventions: Dietary Supplement: Sucrose; Device: Wear smart underwear
- Experimental (Experimental): Participants consume lactose and wear the Smart Underwear device
  Interventions: Dietary Supplement: Lactose; Device: Wear smart underwear

INTERVENTIONS:
Dietary Supplement: Lactose — Participants receive lactose to determine whether it changes gut microbial hydrogen production
  Arms: Experimental
Dietary Supplement: Sucrose — Participants will consume sucrose which they will consume as a placebo
  Arms: Placebo
Device: Wear smart underwear — Participants will wear the smart underwear device to measure the microbiome activity index

SUMMARY:
The goal of this Interventional study is to validate the Smart Underwear device's ability to detect lactose intolerance by comparing its results to self-reported symptoms in adult participants aged 18 and above, divided equally between self-reported lactose-tolerant and lactose-intolerant individuals.

The main questions it aims to answer are:

Can the Smart Underwear device reliably measure flatus events after lactose consumption? Does the Microbiome Activity Index differentiate between responses to lactose and sucrose consumption?

Researchers will compare participants consuming lactose (experimental arm) with their results after consuming sucrose (placebo arm) to see if the device detects increased flatus events and higher Microbiome Activity Index values in the lactose arm.

Participants will:

* Follow a low-fiber/low-FODMAP diet for four days.
* Record meals using a food log and a custom smartphone app.
* Wear the Smart Underwear device for 8 hours daily for three days.
* Fast for 12 hours overnight, consume 20 grams of either lactose or sucrose dissolved in water, and continue fasting for an additional 4 hours.
* Fast for 12 hours overnight, consume 20 grams of the carbohydrate they did not consume the first time (lactose or sucrose) dissolved in water, and continue fasting for an additional 4 hours.
* Complete digestive symptom surveys after each carbohydrate intake.

The randomized crossover design ensures that participants consume both lactose and sucrose on separate days, with blinding maintained for both participants and researchers.

ELIGIBILITY:
Inclusion Criteria:

* Has no gastrointestinal disorders
* Not consuming any prescribed medications
* Willing and able to consume sucrose and lactose
* Determined to be lactose tolerant or lactose intolerant after completing an eligibility survey

Exclusion Criteria:

* Younger than 18 years old
* Diagnosed with or suspected to have the following conditions: diabetes, prediabetes, high blood sugar, IBD, SIBO, or a food allergy to sucrose or lactose
* Experience gastrointestinal pain, bloating, or diarrhea when consuming garlic, onions, or leeks
* Routinely experience constipation or painful constipation
* Have ever had an anaphylactic reaction after eating or drinking anything

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-12-05 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Microbiome activity index | 8 hours from consumption of the lactose and sucrose
  The Microbiome Activity Index A high gut microbiome activity is closely correlated with hydrogen gas production, reflected in the increase of both flatus frequency and hydrogen concentration. It is essential to consider these two variables together. The accumulated gas can be expelled in a few high-intensity events or through a series of smaller flatus. Consequently, relying solely on counting flatus or measuring only the sensor output does not provide a complete picture of gut microbiome activity. Additionally, the investigators found that high concentrations of hydrogen in flatus can sometimes saturate the sensor. To address this issue, the investigators discovered that using the absolute value of the sensor signal's first derivative offers a more accurate assessment of flatus intensity. By measuring the rate of change rather than the signal output, the method can reduce the baseline contribution and better identify flatus.

CONTACTS AND LOCATIONS:
Locations (1):
- Bioscience Research Building, College Park, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
The following Individual Participant Data (IPD) will be shared: Microbiome Activity Index measurements from both the sham control and lactose challenge arms, collected via the Smart Underwear device's electrochemical sensor array during the controlled crossover trial. The Microbiome Activity Index reflects the quantified hydrogen gas events exceeding baseline threshold during the monitoring period. The study protocol and informed consent documents will also be made available. The data represents measurements taken over 8-hour periods following oral lactose or sham administration while participants wore the device.
Supporting Information: Study Protocol, ICF